CLINICAL TRIAL: NCT04647578
Title: Physical Fitness Levels in Children and Adolescents With Chronic Inflammatory Bowel Disease (CIBD): Crohn's Disease, Ulcerative Colitis, Chronic Unclassified Colitis
Acronym: MICI-FIT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Lille (Other)
Collaborators: Groupement Interrégional de Recherche Clinique et d'Innovation (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_03; 2019-A02651-56 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-11-24; First posted 2020-12-01 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Crohn's Enteritis; Crohn Disease; Inflammatory Bowel Diseases; Colitis, Ulcerative; Granulomatous Enteritis; Granulomatous Colitis; Ileocolitis; Proctocolitis
Keywords: Pediatric; IBD; physical fitness
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Colitis, Ulcerative; Proctocolitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Child with IBD
  Interventions: Device: GT3X Actigraph accelerometer.
- Healthy child witnesses

INTERVENTIONS:
Device: GT3X Actigraph accelerometer. — GT3X Actigraph accelerometer during 7 days
  Groups: Child with IBD

SUMMARY:
Inflammatory bowel diseases (IBDs), including Crohn's disease (CD), ulcerative colitis (UC) and IBD-unclassified (IBD-U), are characterised by chronic inflammation of the gastrointestinal tract. Over the past 50 years, the incidence of IBD has increased globally, with the highest increase in industrialised countries. During the last 25 years, the incidence of IBD has increased dramatically among teenagers in northern France, with an increase of 126% and 156% for CD and UC, respectively.

Physical fitness is a set of attributes related to a person's ability to perform physical activities that require aerobic capacity, endurance, strength or flexibility and is determined by a combination of regular physical activity and genetically inherited ability. Physical fitness, widely recognised as an important health determinant, plays an important role in growth and development. Due to the evidence-based importance of physical fitness for young people's health status, attention should be paid to the assessment of physical fitness at these ages and whatever the health status.

At this time, there is no study on the assessment of physical fitness in IBD pediatric patient.

ELIGIBILITY:
Inclusion Criteria:

* For children with IBD:
* boy or girl aged 10 to 17 years old when signing the consent.
* obtain the consent of participation of the child and the signed inform consent of the two parents or a legal representative.
* Patient benefiting from health care- has IBD (Crohn's disease, ulcerative colitis and unclassified chronic colitis) for at least 6 months.
* Contactable by phone

For healthy controls:

* Patient without IBD
* Boy or girl aged 10 to 17 years old when signing the consent.
* obtain the consent of participation of the child and the signed inform consent of the two parents or a legal representative.
* Patient benefiting from health care

Exclusion Criteria:

* For children with IBD:
* Acute intercurrent events at the time of inclusion which may lead to a decrease in physical fitness and activity, according to the judgment of the investigator (fractures, recent arthritis, ano-perineal lesions, severe dermatological lesions).
* Patients with a disease a mild activity (PCDAI score > 30 for children with Crohn disease and PUCAI > 35 for children with ulcerative colitis.
* Chronic, acute or intermittent diseases (other than IBD) that may lead to a decrease in physical activity (Example: fracture, paralysis, blindness ...).
* Refusal of the child's participation in the protocol.
* Refusal of one of the child's parents to participate in the protocol.
* Participation in another interventional study.
* Pregnant or lactating women.
* Patient under protection of justice.

For healthy controls:

* Chronic, acute or intermittent diseases (other than IBD) that may lead to a decrease in physical fitness and activity (Example: fracture, paralysis, blindness ...).
* Refusal of the child's participation in the protocol.
* Refusal of one of the child's parents to participate in the protocol.
* Participation in another interventional study.
* Pregnant or lactating women.
* Patient under protection of justice.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children and adolescents with IBD (Crohn's disease, ulcerative colitis and chronic ulcerative colitis).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Difference in cardiorespiratory fitness (expressed in ml/kg/min) between children and adolescents with IBD and age-, BMI and sex-matched healthy controls. | At 7 days

SECONDARY OUTCOMES:
Difference in muscular endurance, strength, speed/agility, flexibility, strength between children and adolescents with IBD and age-, BMI and sex-matched healthy controls | Baseline, at 7 days
Disease activity according to PCDAI scores | Baseline, at 7 days
  (Pediatric Crohn Disease Activity Index)
Disease activity according to PUCAI scores | Baseline, at 7 days
  Pediatric Ulcerative Colitis Activity Index
Percentage of IBD children and adolescents with a cardiovascular risk disease | Baseline, at 7 days
Correlation between quality of life and physical fitness in children and adolescent with IBD | Baseline, at 7 days
Correlation between fatigue and physical fitness in children and adolescent with IBD | Baseline, at 7 days
Correlation between daily physical activity and physical fitness in children and adolescent with IBD | Baseline, at 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Dominique TURCK, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Jeanne de Flandre Chu Lille, Lille, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. Data will be made available following the conclusion of the project's period of funding.

REFERENCES:
- [Derived] Vanhelst J, Beghin L, Coopman S, Labreuche J, Djeddi D, Gottrand F, Turck D, Ley D. Physical fitness in children and adolescents with inflammatory bowel disease: protocol for a case-control study. BMJ Open. 2022 Oct 11;12(10):e063403. doi: 10.1136/bmjopen-2022-063403. PMID 36220315